CLINICAL TRIAL: NCT05186701
Title: Effects of Kinesio Taping in Protracted Shoulder Posture: a Randomized Control Trial
Brief Title: Effects of Kinesio Taping in Protracted Shoulder Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00565 Anum Khalid
Record Dates: First submitted 2021-10-07; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Postural; Defect
Keywords: Double square; Kinesio taping; Protracted shoulder posture; Tapeline; Total scapular distance; Rrotracted shoulder posture
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: 68 participants were divided in two groups. Group A got Kinesio taping and conventional treatment while group B got only conventional treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kinesio taping and Conventional Physical Therapy (Experimental): Standardized therapeutic kinesio taping (I shaped with 50-100% tension for 72 hours on both shoulders) along with Conventional Physical Therapy including Thermotherapy, myofacial release, exercise therapy (active isolated unilateral stretching of pectoralis minor muscle and strengthening of shoulder retractors).
  Interventions: Other: Kinesio Tape
- Conventional Physical Therapy (Active Comparator): Thermotherapy, myofacial release, exercise therapy (active isolated unilateral stretching of pectoralis minor muscle and strengthening of shoulder retractors).
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Kinesio Tape — Kinesio tape was applied with mechanical correction technique having I shaped with 50-100% tension for 72 hours on both shoulders in retracted position from the anterior aspect of the acromion to the spinous process of the 10th thoracic vertebra of the both shoulders.
  Conventional Physical; Therapy:
  Thermotherapy (hot pack) applied for 10 minutes. Myofacial release. Active isolated unilateral stretching of pectoralis minor muscle for 30 seconds (3 set × 3 reps/day).
  Strengthening of shoulder retractors (lower trapezius and rhomboids). (3 set × 15 reps/day).
  Participants were asked to do exercises at home on daily basis.
  Arms: Kinesio taping and Conventional Physical Therapy
Other: Conventional Physical Therapy — Conventional Treatment: Hot pack, Myofascial Releaase, Stretching and Strengthening with Theraband
  Arms: Conventional Physical Therapy

SUMMARY:
To determine the effects of kinesio taping in protracted shoulder posture.

DETAILED DESCRIPTION:
Office workers generally adopt slumped sitting posture while working at desk for longer durations. Computer use has rapidly increased from past 30 years in various offices so that employees spend plenty of time using computers. Excessive increase in sustained sitting while using computers lead individuals to faulty postures, such as protracted shoulder posture. Changes in posture are related to modifications in muscular functions which alter position of joints and produce movement impairment.

Protracted shoulder/ forward head posture is one of the most prevalent faulty postures in upper quarter. This posture is associated with forwardly tilted, protracted, internally rotated, elevated and abducted position of scapula along with exaggerated cervical lordosis and upper thoracic spine kyphosis.

Muscle imbalance that occurs in this posture includes tightening of anterior shoulder muscles namely pectoralis minor and major, upper trapezius and serratus anterior and the muscles that become weak are posterior shoulder muscles, middle and lower trapezius and rhomboids. This uncoordinated muscle work causes change in scapular kinematics and orientation of glenohumeral complex that further leads to pain in neck, shoulder and arms. The scapulohumeral rhythm disturbs due to the forward shifting of shoulder joint.

Length of pectoralis minor and inadequate strength of lower trapezius are considered to be the vital muscular elements causing protracted shoulder posture in literature review. Tightening of the pectoralis minor is one of the significant feature to cause this posture. This muscle is found to be required for lengthening in individuals having protracted shoulder posture. 78% of variance in this posture was accounted by pectoralis minor muscle.

Protracted shoulder posture is a multifactorial condition and have several treatment protocols including exercises that involves lengthening of hyperactive muscles, strengthening of weak muscles, scapular posterior tilting exercises, massage, bracing or taping, postural correction and soft tissue mobilization.

Kinesio taping is a widely used technique that have ability to stretch longitudinally up to 140-150% of its actual length and was manufactured to replicate the skeletal muscle's elasticity. Depending on direction of pull and percentage of stretch during its application, it provides several benefits i.e it facilitates or inhibit range of motion, gives positional stimulus, produces further space by lifting skin, soft tissues and fascia, provides proper alignment of fascial tissues, decreases pain and edema. The technique which is utilized by clinicians in order to inhibit or facilitate muscles is mechanical correction.

There was limited use of this technique in our society especially for faulty postures and lack of postural awareness in our settings. Current study was planned to examine the effect of Kinesio tape on protracted shoulders.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having bilateral protracted shoulder posture
* Work for at least 7 hours/day, 5 days/week, in a seated position

Exclusion Criteria:

* History of serious pathology (e.g., malignancy, inflammatory disorder, infection)
* History of cervical and thoracic spine and shoulder surgery in previous12 months
* History of trauma or fractures in cervical and thoracic spine
* Any spinal deformities such as Sprengel's deformity, scoliosis, kyphosis etc.
* Diagnosis of psychiatric disorders such as anxiety and depression
* Cervical and thoracic spondylolisthesis, radiculopathy and spinal stenosis
* Severe skin allergy

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Pectoralis Minor Length (PML) | 2nd week.
  Changes from baseline, Pectoralis Minor Length was assessed using tapeline. To determine the pectoralis minor length, distance in inches from the inferior and medial aspect of coracoid process to the inferior edge of fourth rib was taken.
Total Scapular Distance (TSD) | 2nd week.
  Changes from baseline, Total Scapular Distance (TSD) was assessed using tapeline. It was measured by taking distance from third thoracic spinous process to caudal angle of acromion in inches.
Supine measurement of protracted shoulder posture | 2nd week.
  Changes from baseline, Supine measurement of protracted shoulder was measure by Straight ruler which is a simple scale that give measurements in inches or centimeters. Participants lied supine and their arms rested on abdomen with flexed elbows. Then distance was measured from posterolateral aspect of acromion to examining table in inches.
Standing measurement of protracted shoulder posture | 2nd week.
  Changes from baseline, Standing measurement of protracted shoulder posture was mesasure by Double square which is a 12 inches long carpenter square with another square hang over this 12 inch ruler. Participants were asked to stand against wall, this tool was placed parallel to wall over the shoulder to be assessed and positioned it's another extended square at the tip of acromion anteriorly. Then distance from wall to acromion was measured in inches.

CONTACTS AND LOCATIONS:
Overall Officials: Shafaq Shahid, MSPT-OMPT, Principal Investigator — Riphah International University; Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah International University
Locations (1):
- University of Lahore, Islamabad Campus, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No